CLINICAL TRIAL: NCT03975517
Title: Analysis of Sexual Risks in Prep (Pre-exposure Prophylaxis) Users Followed-up in a University Care Centre (Le Trait d'Union)
Brief Title: Sexual Risks in Prep Users
Acronym: PREP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7300
Record Dates: First submitted 2019-03-18; First posted 2019-06-05 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: HIV Infection; Prep Prescription; Vaccinations; Sexually Transmitted Diseases
Keywords: Prep; Sexual behavior; HIV; Syphilis; Chlamydia infection; Hepatitis; Gonococcus
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Sexual Behavior; Syphilis; Chlamydia Infections; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: PrEP — Define the behavioral characteristics of the active file of patients using PrEP in Strasbourg in 2019.

SUMMARY:
Primary purpose of the study: to describe sexual behavior of Prep users, whatever mode of intake, ie continuous or on-demand; it has been shown in some studies, an increase of sexual risks in Prep users, and therefore an similar increase of STIs (sexually transmitted diseases); using a self-questionnaire, we'd like to evaluate sexual behavior before, and 6 months after, starting Prep.

Secondary purposes: to describe medical characteristics of Prep users (past medical condition, demographic characteristics, vaccinations, kidney function, serological results, urine and anal/pharyngeal swabs), clinical and biological Prep safety, STIs occurrence, and antibiotic prescriptions, continuous or on-demand intake, Prep indication.

ELIGIBILITY:
Inclusion Criteria:

* non HIV-infected subjects
* men aged 18 years or older
* having non protected sexual relationship
* taking Prep (emtricitable/tenofovir disoproxil fumarate) either every day, or on-demand
* affiliated to social security

Exclusion criteria:

* HIV-infected patients
* refusal of study participation
* not on Prep
* not fluent in French language
* safeguarding justice
* on guardianship or trusteeship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non HIV-infected subjects, who have a high risk to be infected by HIV, mostly because of non protected sexual intercourse.
  Most of them are MSM (men who have sex with men). And who started Prep (emtricitable/tenofovir disoproxil fumarate), or will initiate Prep
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Analysis of sexual behavior in Prep users | 6 months
  Sexual behavior will be evaluated with a questionnaire

SECONDARY OUTCOMES:
Description of the medical profile of the Strasbourgeoise active file | 6 months
  Describe the active line of people using Prep and followed in the center

CONTACTS AND LOCATIONS:
Overall Officials: David REY, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided